CLINICAL TRIAL: NCT01669642
Title: Mean Effective Dose of Rapidly Administered Ketamine for Brief Pediatric Procedural Sedation
Brief Title: Study to Find the Dose of Rapidly Administered Ketamine for Brief Painful Procedures in Children
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Washington University School of Medicine (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 201112017
Record Dates: First submitted 2012-08-08; First posted 2012-08-21 (Estimated); Results first posted 2018-03-12 (Actual); Last update posted 2019-04-25 (Actual); Status verified 2019-04

CONDITIONS: Abscess; Fracture
Keywords: ketamine sedation; pediatric; abscess drainage; fracture reduction
MeSH Terms: conditions — Abscess; Fractures, Bone | interventions — Ketamine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Ketamine (Experimental): participants who get the ketamine sedation will be enrolled. there is no control or comparison group.
  Interventions: Drug: Ketamine

INTERVENTIONS:
Drug: Ketamine — participants who need ketamine sedation for abscess drainage or fracture reduction will be approached for enrollment. there is no comparison group. A predetermined dose of Ketamine will be administered over 5 seconds or less intravenously. Sedation provider will assess for effectiveness of sedation at one minute.
  Other Names: Ketalar

SUMMARY:
The purpose of the study is to find the dose of rapidly administered ketamine in 3 different pediatric age groups (2-5, 6-11 and 12-17) for abscess drainage and fracture reduction.

Ketamine is the most common drug administered to children to facilitate painful procedures in the emergency setting because it achieves potent sedation, pain relief and amnesia with minimal adverse cardiopulmonary effects.(1-5) However, the 1-2 hour recovery period (1,6) associated with standard ketamine administration guidelines(7) strains work flow because it requires bedside one-on-one nurse monitoring in a treatment room, tying up these limited and valuable resources. Consequently, a combination of two other drugs, propofol + fentanyl (P/F), with recovery of 20-30 minutes, is rapidly gaining popularity for procedural sedation despite more frequent respiratory depression, apnea and hypotension caused by this technique.(2,4,8,9)

The investigators believe recovery associated with our novel method for administering ketamine is significantly shorter than with the standard larger dose more slowly administered ketamine technique(7). Through the investigators clinical experience, the investigators have found rapid infusion of smaller than standard doses of ketamine safely achieves the drug's sedative effect, with the benefit of more rapid recovery due to the use of a smaller dose. However, this novel technique challenges published beliefs that time of recovery from ketamine sedation does not differ significantly with the dose administered, within the usual dose ranges, and that rapid infusion may cause respiratory depression, similar to that seen with other classes of sedative-analgesic drugs.(7,10) the investigators believe the slow infusion recommended by standard guidelines(7) requires a larger ketamine dose necessary to achieve effective sedation, and, consequently, prolongs recovery. It is the prolonged recovery that has prompted increased use of other less safe but briefer sedatives, such as propofol/fentanyl. By demonstrating patients recover rapidly with new ketamine technique, without increased adverse cardiopulmonary effects, the investigators will provide clinicians with an important new method for ketamine procedural sedation. The investigators believe clinicians will prefer more rapid recovery ketamine technique because it is safer and reduces pain and distress better than the propofol/fentanyl combination for sedation.

The investigators complete proposal requires two steps. In Step One, this proposal, the investigators will determine the minimum effective dose of rapidly infused ketamine that achieves deep sedation for at least 5 minutes in 95% of children (ED95). Two groups of patients will be studied: one group is patients undergoing abscess incision and drainage and the other group is patients undergoing fracture reduction in our Emergency Department. The investigators believe that the ED95 is different for both the groups as the severity of pain is different. The investigators will compare the safety and recovery times to published standard ketamine techniques. In the following study, Step Two, the investigators will compare this novel technique, in a blinded randomized trial using the ED95 ketamine dose determined in Step One to the standard ketamine technique to determine if the novel technique results in significantly shorter recovery without an increase in the frequency of adverse effects. The study the investigators are proposing in this submission is Step One only.

DETAILED DESCRIPTION:
During fracture reduction in children, the investigators found less distress using ketamine+midazolam (K/M) sedation (P<0.0001) and less hypoxia (5% vs. 25%) compared to sedation with fentanyl+midazolam (F/M)(1). Others also found less hypoxia with K/M (4%) compared to propofol+fentanyl (P/F) (18-31%)(2,4). Because of the greater safety and efficacy determined in these and similar studies, ketamine is now the most common drug administered for procedural sedation of children undergoing painful procedures in the ED.(7) For the past 15 years, the investigators have sedated about 2,500 children each year with ketamine in the St. Louis Children's Emergency Department for setting broken bones, debriding burns, draining abscesses, and other very painful procedures. Midazolam was co-administered with ketamine in early studies to reduce dysphoria during recovery, but this practice has since been shown not to be beneficial. For the past 5-10 years the investigators have used ketamine without midazolam and have seen no change in how children wake up from ketamine sedation.(6,11)

Ketamine administration in the investigators previous studies (1,3) was similar to recent recommendations (1.5-2 mg/kg I.V. infused over 30-60 sec)(7). Problematically, while most of these ED procedures such as fracture reduction, burn debridement, or abscess incision and drainage, require only 5-10 minutes of deep sedation, this standard ketamine technique results in recovery periods of 60-120 minutes(1,3,6). During recovery, patients remain in treatment rooms to be monitored one-on-one by nurses for respiratory depression, airway obstruction, vomiting and other potentially life-threatening adverse events, thus tying up these limited resources(10). This long recovery has led to increased use of propofol based techniques which have more rapid recovery (20-30 minutes) but cause increased respiratory depression and hypotension and less effective sedation(2-6,9). Because of ketamine's greater safety and efficacy profile, the investigators have been interested in developing alternative ketamine administration regimens that result in more rapid recovery, similar to propofol. If successful in hastening recovery, the investigators believe that the relative lack of respiratory depression and greater analgesia with ketamine will improve patient safety by encouraging continued use of ketamine as the preferred technique for procedural sedation in children undergoing painful procedures in the ED.

To explore new techniques for hastening recovery from sedation, the investigators took advantage of the uniqueness of ketamine. Rapid administration of opioid and gabaergic drugs such as fentanyl and propofol significantly augments the drugs' beneficial effects, but it also markedly increases respiratory depression, apnea and hypotension.(13) Cautions that rapid infusion of ketamine may cause brief respiratory depression stem from early anesthesia trials using doses larger than those typically used for sedation.(7) Although not formally studied, for the past 5 years the investigators have observed no adverse effects with rapid administration of 0.5-1.5 mg/kg ketamine doses for brief painful procedures like fracture reduction and abscess incision & drainage in children in the Emergency Unit of St. Louis Children's Hospital.

Lipophilic drugs used for procedural sedation-analgesia, such as ketamine, fentanyl, and propofol rapidly diffuse from the bloodstream into the brain. A disproportionately high percentage of the cardiac output goes to the brain, thus a large portion of a drug injected intravenously initially goes into the brain's circulation on first pass through the heart and exerts clinical effects within a single circulation time, usually < 60 seconds. The drug remaining in the bloodstream circulates throughout the body and diffuses into muscle, bone and fat, causing the blood concentration to fall. The blood-brain concentration gradient then favors drug diffusion out of the brain and the patient awakens.

Rapid infusion of sedative drugs increases central nervous system clinical effects by directing a larger portion of the drug into the brain. A rapidly injected dose of drug travels as a more concentrated bolus into the brain circulation than a slowly injected dose that is diluted by the passing blood. With rapid injection, therefore, the initial blood-brain concentration gradient is greater and a larger portion of the dose initially enters the brain, causing deeper sedation. Smaller doses, rapidly injected, therefore can be used to achieve deep sedation similar to that of larger doses injected more slowly. With the smaller dose, the blood-brain concentration gradient subsequently reverses more rapidly and "wake up time" is shorter. Because rapid increases in brain concentration of ketamine does not cause respiratory depression, unlike that seen with fentanyl or propofol, this rapid infusion technique can be used with ketamine.

The purpose of this research project is to determine formally the minimum dose of ketamine that, when rapidly infused, achieves 5 minutes of deep sedation in 95% of patients (ED95). The investigators will use the up and down method (15) which is a standard method in anesthesiology to find the mean effective dose. Five minutes is typically enough time to perform these brief painful procedures. The investigators anticipate the ED95 will be smaller than the standard recommended ketamine dose and thus patients will wake up faster.

Of special note, determination of the "standard dose and rate of administration of ketamine"(7) has been based upon our and others' studies in which the dose and rate of infusion of ketamine were not carefully controlled and, in fact, varied widely(1,3,4,7). Thus, the "standard recommendation for administration of ketamine" is somewhat anecdotal and has not been precisely determined. Our proposed study will be the first to precisely determine a minimum effective ketamine dose.

ELIGIBILITY:
Inclusion Criteria:

Healthy children (ASA Physical Status I and II) 2-17 yrs old who require deep sedation for abscess incision and drainage in the St. Louis Children's Hospital Emergency Unit

Exclusion Criteria:

1. Fever (temperature ≥ 38 0Celcius) due to upper respiratory infection.
2. Obesity (BMI > 2SD for age and sex) or undernourishment (BMI < 2SD for age and sex)
3. Children with psychosis/psychiatric diagnosis (currently under the care of psychiatrist and/or taking psychiatric medication. ADHD is not an exclusion criterion)
4. Previous adverse reactions with ketamine sedation
5. Receipt of opioid analgesic in the ED (oxycodone/morphine etc) prior to sedation
6. Multiple abscesses (2 or more) requiring I & D
7. Non -English speaking families
8. Children under foster care.
9. Previous participation in current research study

Ages: 2 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 111 (Actual)
Dates: Start 2012-04; Primary Completion 2014-08 (Actual); Study Completion 2014-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: sri s chinta, MD, Principal Investigator — Washington University School of Medicine
Locations (1):
- St Louis Children's hospital, Washington university, St Louis, Missouri, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: children between 2-18 years of age who presented to st louis children's hospital emergency department between april 2012 and august 2014 with a fracture that needed reduction or a skin abscess that needed drainage under sedation were approached for enrollment.
Groups:
- Fracture Reduction Group 2-5 Years: children between 2-5 years who needs ketamine sedation for fracture reduction in the emergency department are enrolled in this group.
- Fracture Reduction Group 6-11 Years: children between 6-11 years who needs ketamine sedation for fracture reduction in the emergency department are enrolled in this group.
- Fracture Reduction Group 12-17 Years: children between 12-17 years who needs ketamine sedation for fracture reduction in the emergency department are enrolled in this group.
- Abscess Drainage Group 2-5 Years: children between 2-5 years who needs ketamine sedation for abscess drainage in the emergency department are enrolled in this group.
- Abscess Drainage Group 6-11 Years: children between 6-11 years who needs ketamine sedation for abscess drainage in the emergency department are enrolled in this group.
- Abscess Drainage Group 12-17 Years: children between 12-17 years who needs ketamine sedation for abscess drainage in the emergency department are enrolled in this group.
Period: Overall Study
Arm/Group | Fracture Reduction Group 2-5 Years | Fracture Reduction Group 6-11 Years | Fracture Reduction Group 12-17 Years | Abscess Drainage Group 2-5 Years | Abscess Drainage Group 6-11 Years | Abscess Drainage Group 12-17 Years
Started | 20 | 20 | 20 | 21 | 20 | 10
Completed | 20 | 20 | 20 | 20 | 20 | 0
Not Completed | 0 | 0 | 0 | 1 | 0 | 10

BASELINE CHARACTERISTICS:
Groups:
- Fracture Reduction Group 2-5 Years; Fracture Reduction Group 6-11 Years; Fracture Reduction Group 12-17 Years: participants who need ketamine sedation for fracture reduction will be approached for enrollment. A predetermined dose of Ketamine will be administered over 5 seconds or less intravenously. Sedation provider will assess for effectiveness of sedation at one minute.
- Abscess Drainage Group 2-5 Years; Abscess Drainage Group 6-11 Years: participants who need ketamine sedation for abscess drainage will be approached for enrollment. A predetermined dose of Ketamine will be administered over 5 seconds or less intravenously. Sedation provider will assess for effectiveness of sedation at one minute.
- Total: Total of all reporting groups
Arm/Group | Fracture Reduction Group 2-5 Years | Fracture Reduction Group 6-11 Years | Fracture Reduction Group 12-17 Years | Abscess Drainage Group 2-5 Years | Abscess Drainage Group 6-11 Years | Total
Number analyzed (Participants) | 20 | 20 | 20 | 20 | 20 | 100
Age, Continuous [Median (Full Range); unit: years] | 4.8 [2.9 to 5.9] | 9.2 [6 to 11.9] | 13.7 [12.6 to 16.9] | 2.9 [2 to 5.1] | 7.2 [6.4 to 11.9] | 7.2 [2.9 to 11.9]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9 | 6 | 1 | 8 | 11 | 35
  Male | 11 | 14 | 19 | 12 | 9 | 65
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  african american | 5 | 2 | 8 | 9 | 8 | 32
  Caucasian | 13 | 1 | 2 | 10 | 12 | 38
  other | 2 | 17 | 10 | 1 | 0 | 30
Patients who received Opioids prior to sedation [Count of Participants; unit: Participants] | 19 | 18 | 19 | 0 | 0 | 56
time between opioid administration and sedation start time [Median (Full Range); unit: minutes] | 116 [20 to 383] | 96 [1 to 251] | 129 [27 to 401] | 0 [0 to 0] | 0 [0 to 0] | 116 [1 to 401]
fracture characteristics [Count of Participants; unit: Participants]
  Non displaced fracture | 10 | 2 | 9 | 0 | 0 | 21
  displaced fracture but not overriding | 6 | 11 | 7 | 0 | 0 | 24
  displaced fracture and overriding | 4 | 7 | 4 | 0 | 0 | 15
  no fracture | 0 | 0 | 0 | 20 | 20 | 40

OUTCOME MEASURES:

1. Primary Outcome: Median Effective Dose (ED50) and ED95 of Rapidly Administered Ketamine
Description: ED50 is the dose of rapidly administered ketamine that achieves effective sedation in 50% of patients. ED95 is the dose of ketamine that can provide effective sedation in 95% of children undergoing abscess drainage or fracture reduction. ED95 will be calculated for the 3 age groups (2-5, 6-11 and 12-17) independently for both the procedures: abscess drainage and fracture reduction.
Time Frame: Dose administration through 5 minutes
Population: 100 children were enrolled in 5 different groups depending on the age and type of procedure.
Measure: Median (Full Range); unit: mg/kg of ketamine dose
Groups:
- Fracture Reduction Group 2-5 Years: children between 2-5 years of age who need fracture reduction under ketamine sedation are enrolled in this group.
- Fracture Reduction Group 6-11 Years: children between 6-11 years of age who need fracture reduction under ketamine sedation are enrolled in this group.
- Fracture Reduction Group 12-17 Years: children between 12-17 years of age who need fracture reduction under ketamine sedation are enrolled in this group.
- Abscess Drainage Group 2-5 Years: children between 2-5 years of age who need abscess drainage under ketamine sedation are enrolled in this group.
- Abscess Drainage Group 6-11 Years: children between 6-11 years of age who need abscess drainage under ketamine sedation are enrolled in this group.
Arm/Group | Fracture Reduction Group 2-5 Years | Fracture Reduction Group 6-11 Years | Fracture Reduction Group 12-17 Years | Abscess Drainage Group 2-5 Years | Abscess Drainage Group 6-11 Years
Number analyzed (Participants) | 20 | 20 | 20 | 20 | 20
mg/kg of ketamine dose | 0.7 [0.6 to 0.9] | 0.5 [0.5 to 0.7] | 0.6 [0.5 to 0.8] | 0.9 [0.7 to 1.1] | 0.6 [0.4 to 0.9]

2. Primary Outcome: ED95
Description: ED95 is the dose of ketamine effective for 95% of children. this outcome is estimated from ED50.
Time Frame: Dose administration through 5 minutes
Measure: Number; unit: mg/kg of ketamine dose
Arm/Group | Fracture Reduction Group 2-5 Years | Fracture Reduction Group 6-11 Years | Fracture Reduction Group 12-17 Years | Abscess Drainage Group 2-5 Years | Abscess Drainage Group 6-11 Years
Number analyzed (Participants) | 20 | 20 | 20 | 20 | 20
mg/kg of ketamine dose | 0.7 | 0.7 | 0.8 | 1.1 | 1.1

3. Secondary Outcome: Vomiting
Description: patients who experienced vomiting while in the ED or after discharge
Time Frame: Administration of ketamine through 2 week follow up call
Measure: Count of Participants; unit: Participants
Arm/Group | Fracture Reduction Group 2-5 Years | Fracture Reduction Group 6-11 Years | Fracture Reduction Group 12-17 Years | Abscess Drainage Group 2-5 Years | Abscess Drainage Group 6-11 Years
Number analyzed (Participants) | 20 | 20 | 20 | 20 | 20
Participants
  vomiting in the ED | 1 | 1 | 1 | 1 | 0
  Vomiting after discharge | 6 | 3 | 3 | 2 | 1
  No vomiting | 13 | 16 | 16 | 17 | 19

4. Secondary Outcome: Number of Participants With Wisconsin Sedation Scale Score of 2 or Less at 1 Minute After First Dose of Ketamine
Description: This is a measure of sedation effectiveness; to assess the effectiveness of first dose of ketamine administered.
  Possible values for the scale range from 0 to 6. A sedation score of 2 or less is considered adequate sedation. Values more than 2 indicate state of inadequate sedation. higher values indicate the need for additional doses of sedation.
  Patients who achieved a score of 2 or less are considered effective sedation and a score of >2 are considered ineffective sedations.
Time Frame: Dose administration through 1 minute
Measure: Number; unit: participants
Arm/Group | Fracture Reduction Group 2-5 Years | Fracture Reduction Group 6-11 Years | Fracture Reduction Group 12-17 Years | Abscess Drainage Group 2-5 Years | Abscess Drainage Group 6-11 Years
Number analyzed (Participants) | 20 | 20 | 20 | 20 | 20
participants | 12 | 9 | 10 | 13 | 10

5. Other Pre Specified Outcome: Total Sedation Time
Description: during recovery, all participants are monitored for recovery to baseline at which point participants are ready for discharge. we will document the time from induction to recovery to aldrete score of 10.
Time Frame: Time of administration of ketamine through sedation recovery
Measure: Median (Full Range); unit: minutes
Arm/Group | Fracture Reduction Group 2-5 Years | Fracture Reduction Group 6-11 Years | Fracture Reduction Group 12-17 Years | Abscess Drainage Group 2-5 Years | Abscess Drainage Group 6-11 Years
Number analyzed (Participants) | 20 | 20 | 20 | 20 | 20
minutes
  Patients requiring single dose of ketamine | 25 [15 to 30] | 22.5 [15 to 31] | 25 [25 to 30] | 20.5 [13 to 40] | 17.5 [10 to 40]
  patients requiring more than single dose | 35 [25 to 85] | 25 [15 to 50] | 45 [20 to 80] | 27.5 [16 to 40] | 35 [10 to 60]

ADVERSE EVENTS:
Time Frame: from the day of enrollment up to 2 weeks.
Arm/Group | Fracture Reduction Group 2-5 Years | Fracture Reduction Group 6-11 Years | Fracture Reduction Group 12-17 Years | Abscess Drainage Group 2-5 Years | Abscess Drainage Group 6-11 Years
All-Cause Mortality (participants affected / at risk) | 0/20 | 0/20 | 0/20 | 0/20 | 0/20
Serious Adverse Events (participants affected / at risk) | 0/20 | 0/20 | 0/20 | 0/20 | 0/20
Other Adverse Events (participants affected / at risk) | 7/20 | 5/20 | 7/20 | 3/20 | 2/20
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Fracture Reduction Group 2-5 Years (N=20) | Fracture Reduction Group 6-11 Years (N=20) | Fracture Reduction Group 12-17 Years (N=20) | Abscess Drainage Group 2-5 Years (N=20) | Abscess Drainage Group 6-11 Years (N=20)
dysphoria, ag (Nervous system disorders) | 0 (0) | 1 (1) | 3 (3) | 0 (0) | 1 (1) — patients who experienced dysphoria during sedation or recovery period
vomiting (Gastrointestinal disorders) | 7 (7) | 4 (4) | 4 (4) | 3 (3) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes